CLINICAL TRIAL: NCT06696261
Title: A Multicenter, Randomized, Double-blind, Placebo Parallel-controlled Phase III Clinical Trial on the Efficacy and Safety of Lianxiaxiaopi Granules in the Treatment of Postprandial Distress Syndrome (Intermingled Cold and Heat).
Brief Title: A Study of Lianxiaxiaopi Granules in the Treatment of Postprandial Distress Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-LXXPKL-Ⅲ
Record Dates: First submitted 2024-11-08; First posted 2024-11-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postprandial Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lianxiaxiaopi Granules (Experimental)
  Interventions: Drug: Lianxiaxiaopi Granules
- a simulated agent of Lianxiaxiaopi Granules (Placebo Comparator)
  Interventions: Drug: a simulated agent of Lianxiaxiaopi Granules

INTERVENTIONS:
Drug: Lianxiaxiaopi Granules — The participants took orally 1 sachet of Lianxiaxiaopi Granules, 3 times a day for 8 weeks.
  Arms: Lianxiaxiaopi Granules
Drug: a simulated agent of Lianxiaxiaopi Granules — The participants took orally 1 sachet of simulated agent of Lianxiaxiaopi Granules, 3 times a day for 8 weeks.
  Arms: a simulated agent of Lianxiaxiaopi Granules

SUMMARY:
The goal of this clinical trial is evaluating the efficacy and safety of Lianxiaxiaopi Granules in participant population. The main questions it aims to answer are:

1. Based on the Response rate of postprandial distress syndrome participants, evaluate whether the efficacy of Lianxiaxiaopi Granules is superior to placebo.
2. Evaluate the efficacy of Lianxiaxiaopi Granules in improving symptom of postprandial distress syndrome.
3. Evaluating the safety of Lianxiaxiaopi Granules in postprandial distress syndrome participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years old (including boundary value), gender is not limited;
2. meet the diagnostic criteria for postprandial distress syndrome (Rome IV.);
3. Meet the syndrome differentiation standards of Traditional Chinese Medicine for cold and heat miscellaneous syndromes;
4. NRS score of at least one symptom of postprandial distress syndrome (postprandial fullness, discomfort, early satiety) in the screening period and baseline period≥ 4 points; and did not have moderate/severe epigastric pain syndrome (mid-epigastric burning sensation and mid-upper quadrant pain both < 4 points);
5. Those who did not have organic abnormal changes in the results of gastroscopy (including no abnormalities in gastroscopy, chronic non-atrophic gastritis/chronic superficial gastritis with erythema grade I and/or erosion that was flat and only grade I);
6. Negative Helicobacter pylori test in 13C/14C breath test during the screening period;
7. Voluntarily participate in clinical trials, sign informed consent, and understand and comply with research procedures.

Exclusion Criteria:

1. Those who have undergone Helicobacter pylori eradication treatment within 6 months before screening;
2. Gastric mucosal erythema grade II or above, erosion is bulge or grade II or above, or accompanied by bleeding, bile reflux, ≥ 3 inflammatory polyps and other manifestations, or combined with pathological diagnosis of chronic atrophic gastritis, hyperplastic polyps, glandular polyps, etc.; or those who have been clearly diagnosed with dyspepsia caused by organic diseases of the digestive system, such as digestive tract tumors, hepatobiliary and pancreatic diseases, inflammatory bowel diseases, etc.; or those who have other diseases that affect the evaluation of dyspepsia-related symptoms in the past, such as reflux esophagitis, peptic ulcer, gastrointestinal bleeding, intestinal obstruction, etc.;
3. Those who have been diagnosed with systemic diseases that seriously affect the function of the digestive tract, such as hyperthyroidism or hypothyroidism, diabetes, chronic renal insufficiency, connective tissue diseases, etc.;
4. Patients with severe cardiovascular and cerebrovascular, liver, lung, kidney, blood or systemic diseases that affect their survival; or patients with severe mental illness in the past, such as moderate or severe depression/anxiety/bipolar disorder, etc.;
5. Those who have a history of major abdominal surgery in the past, which may affect gastrointestinal function (except for appendectomy, cesarean section, endoscopic colon polyp resection and other surgeries that do not affect digestive function);
6. Patients with abnormal liver function (ALT or AST >1.5 times the upper limit of normal) or abnormal renal function test (Cr> upper limit of normal);
7. Glycosylated hemoglobin ≥ 6.5% or fasting blood glucose ≥7mmol/L during the screening period;
8. Use of drugs or treatments that may have an impact on the effectiveness assessment of the trial drug within 2 weeks before screening (such as acid/antacids, gastrointestinal motility drugs, digestive enzymes, gastric mucosal protectors, antiemetics, antispasmodics, macrolide antimicrobials, azole antifungals, non-steroidal anti-inflammatory drugs, glucocorticoids, anti-anxiety and depressants, analgesics, sedatives; as well as traditional Chinese medicine decoctions, proprietary Chinese medicines and acupuncture treatments for the treatment of functional dyspepsia, etc.);
9. Pregnant and lactating women, who have a birth plan within one month after enrollment and the end of the trial;
10. Those who suspect or have a history of alcohol or drug abuse;
11. Participated in other clinical trials within 1 month before screening;
12. Those who are suspected or known to be allergic to the ingredients of this medicine;
13. According to the judgment of the investigator, it is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial distress syndrome response rate | The end of Week 8
  Postprandial Distress Syndrome Response, the number of weeks in which the subject responded to the postprandial distress syndrome was greater than 50% of the weeks throughout the treatment period.
  Response week, if the two symptoms of postprandial fullness and discomfort and early satiety decreased by ≥50% compared with the baseline per week, the response week was calculated by the diary card score.

SECONDARY OUTCOMES:
postprandial distress syndrome score change from baseline | The end of Week 8
  "The dyspepsia symptom scoring criteria" consists of 5 items, with a minimum score of 0 and a maximum of 10 points for each item.
  0 points: asymptomatic; 1-3 points: mild disturbance, mild symptoms, almost no impact on daily life and work; 4-6 points: moderate disturbance, still tolerable, partially affecting daily life and work; 7-10 points: Severe disturbance, unbearable, unable to carry out daily life and work.
  The minimum score of the scale is 0 points, the maximum is 50 points, and the higher the score, the more serious the disease.
single symptom response rate | The end of Week 8
the change value of single symptom score from baseline | The end of Week 8
  "The dyspepsia symptom scoring criteria" consists of 5 items, with a minimum score of 0 and a maximum of 10 points for each item.
  0 points: asymptomatic; 1-3 points: mild disturbance, mild symptoms, almost no impact on daily life and work; 4-6 points: moderate disturbance, still tolerable, partially affecting daily life and work; 7-10 points: Severe disturbance, unbearable, unable to carry out daily life and work.
the change from baseline in epigstric pain syndrome score | The end of Week 8
  "The dyspepsia symptom scoring criteria" consists of 5 items, with a minimum score of 0 and a maximum of 10 points for each item.
  0 points: asymptomatic; 1-3 points: mild disturbance, mild symptoms, almost no impact on daily life and work; 4-6 points: moderate disturbance, still tolerable, partially affecting daily life and work; 7-10 points: Severe disturbance, unbearable, unable to carry out daily life and work.
  The score for epigastric pain syndrome includes the sum of the scores for mid-upper quadrant pain and mid-upper quadrant burning sensation
epigastric pain syndrome response rate | The end of Week 8
the change from baseline in the total score of TCM | The end of Week 8
  The TCM Syndrome Scale for Postprandial Distress Syndrome contains two main symptoms, each of which can be evaluated as 0, 2, 4 and 6 points. 6 sub-symptoms, each of which can be evaluated as 0, 1, 2, and 3 points.
  The scale has a minimum score of 0 and a maximum of 30 points, with the higher the score, the more severe the condition.
the change value of TCM single symptom score from baseline | The end of Week 8
  The TCM Syndrome Scale for Postprandial Distress Syndrome contains two main symptoms, each of which can be evaluated as 0, 2, 4 and 6 points. 6 sub-symptoms, each of which can be evaluated as 0, 1, 2, and 3 points.
  The scale has a minimum score of 0 and a maximum of 30 points, with the higher the score, the more severe the condition.
TCM syndrome integral effective rate | The end of Week 8
  Recovery: Symptoms and signs disappear or basically disappear, and the score reduction rate of the syndrome ≥95%; Effective: Symptoms and signs improved, and the score reduction rate of the syndrome was ≥50%; Ineffective: no significant improvement in symptoms and signs, and the score reduction rate of the syndrome <50%.
  Recovery: Symptoms and signs disappear or basically disappear, and the score reduction rate of the syndrome ≥95%; Effective: Symptoms and signs improved, and the score reduction rate of the syndrome was ≥50%; Ineffective: no significant improvement in symptoms and signs, and the score reduction rate of the syndrome <50%.
  Recovery: Symptoms and signs disappear or basically disappear, and the score reduction rate of the syndrome ≥95%; Effective: Symptoms and signs improved, and the score reduction rate of the syndrome was ≥50%; Ineffective: no significant improvement in symptoms and signs, and the score reduction rate of the syndrome <50%.
the grade change of TCM single symptom from baseline | The end of Week 8
  The TCM Syndrome Scale for Postprandial Distress Syndrome contains two main symptoms, each of which can be evaluated as 0, 2, 4 and 6 points. 6 sub-symptoms, each of which can be evaluated as 0, 1, 2, and 3 points.
  The scale has a minimum score of 0 and a maximum of 30 points, with the higher the score, the more severe the condition.
the proportion of subjects with sustained remission and no exacerbation of single symptoms at 12W compared with 8W | The end of Week 12
  There are 5 items in the Likert scale, with a minimum score of 1 and a maximum of 7 points for each item. The scale has a minimum score of 0 and a maximum of 35 points, with higher scores and more severe conditions.
  Among them, the subjects selected (1) and (2) are defined as having sustained remission from treatment; Subjects selected (3) and (4) were defined as having no exacerbation of disease; Subjects selected (5), (6), and (7) were defined as having exacerbated disease.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou, Gansu
  - The First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine, Guiyang, Guizhou
  - Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Baoding No. 1 Hospital of Traditional Chinese Medicine, Baoding, Heibei
  - The First People's Hospital of Luoyang City, Luoyang, Henan
  - The Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin
  - General Hospital of the Northern Theater of the Chinese People's Liberation Army, Shenyang, Liaoning
  - The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Shaanxi University of Traditional Chinese Medicine, Xianyang, Shanxi
  - The Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou, Zhejiang